CLINICAL TRIAL: NCT06750003
Title: 4K Versus 3D Total Laparoscopic Bilateral Oophorectomy by Surgeons in Training: Tools in Comparison
Brief Title: 4K Versus 3D Total Laparoscopic Bilateral Oophorectomy: Tools in Comparison
Acronym: TOLSTOY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Stefano Restaino, Doctor, Azienda Sanitaria-Universitaria Integrata di Udine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33935
Record Dates: First submitted 2024-12-15; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Diseases
Keywords: Benign ovarian disease; laparoscopy; annessiectomy; ovariectomy; resident; tridimensional; high definition surgery; 3D; 4K
MeSH Terms: conditions — Ovarian Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D laparoscopy (Active Comparator): Performed using 3D laparoscopy
  Interventions: Procedure: 3D versus 4K laparoscopic bilateral salpingo-oophorectomy
- 4K laparoscopy (Experimental): Performed using 4K laparoscopy
  Interventions: Procedure: 3D versus 4K laparoscopic bilateral salpingo-oophorectomy

INTERVENTIONS:
Procedure: 3D versus 4K laparoscopic bilateral salpingo-oophorectomy — 3D laparoscopy versus 4K laparoscopy for bilateral salpingo-oophorectomy performed by residents

SUMMARY:
Evaluate whether the 4K laparoscopic vision system can provide an advantage in performing bilateral oophorectomy procedures for benign conditions carried out by trainee surgeons compared to 3D laparoscopy

DETAILED DESCRIPTION:
All patients diagnosed with suspected benign ovarian pathology based on preoperative examinations (pelvic Doppler ultrasound and/or magnetic resonance imaging and/or CT scan) and with indication for bilateral laparoscopic adnexectomy will be enrolled in the study. The primary objective of the study is to compare surgical times between the 3D and 4K vision systems in laparoscopic ovarian surgery, specifically in bilateral adnexectomy performed by trainee surgeons. Secondary objectives will include evaluating intra- and postoperative complications, length of hospital stay, and costs to the healthcare system

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign ovarian pathology requiring bilateral oophorectomy
* ASA score <3
* Patients who have signed the appropriate informed consent
* Patients who are not pregnant or diagnosed with pelvic inflammatory disease
* No history of prior major abdominal surgery

Exclusion Criteria:

* Suspected neoplastic pathology
* Patients not eligible for surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
operative time | from enrollment to the end of follow up at 12 months
  To compare the operative time of bilateral oophorectomy performed using 3D laparoscopy versus 4K laparoscopy for benign indications, conducted by trainee surgeons.

IPD SHARING:
Plan to Share IPD: No